CLINICAL TRIAL: NCT02330289
Title: The Effect of Norms on Laboratory and Imaging Testing (ENLITen): a Pragmatic Randomized Controlled Trial
Brief Title: Effect of Norms on Laboratory and Imaging Testing (ENLITen)
Acronym: ENLITen
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Principal Investigator, Kira Ryskina, Fellow, Division of General Internal Medicine, University of Pennsylvania
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 820924
Record Dates: First submitted 2014-12-29; First posted 2015-01-01 (Estimated); Last update posted 2023-04-06 (Actual); Status verified 2023-04

CONDITIONS: Utilization; Laboratory, Hospital
MeSH Terms: conditions — Patient Acceptance of Health Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Report card arm (Experimental): The intervention arm will receive an email report card describing their lab use compared to their peers as well as a link to a website visually tracking the team's daily ordering of common lab tests compared to the peer teams.
  Interventions: Behavioral: Normative report card
- Control arm (No Intervention): Physicians in the control arm will not receive the email or website link.

INTERVENTIONS:
Behavioral: Normative report card — Personalized visual report card describing physician's laboratory ordering pattern for prior week relative to peers as well as a link to a website tracking lab ordering for the team in real time compared to peer teams.
  Arms: Report card arm

SUMMARY:
Studies suggest that some laboratory tests ordered for hospitalized patients are duplicative or have limited value. This study will evaluate a normative feedback intervention to reduce overuse of laboratory tests for hospitalized patients by internal medicine physicians-in-training.

DETAILED DESCRIPTION:
Past research has shown that 25% of diagnostic testing is duplicative or has limited value. Academic medical centers that employ physicians-in-training may find it particularly challenging to reduce low value testing due to a historical emphasis on extensive workups by trainees. Despite the increased emphasis on cost-consciousness in medical education, there is little existing research evaluating ways to optimize ordering behaviors of physicians-in-training. This study will evaluate a normative feedback intervention for internal medicine physicians-in-training to reduce overuse of routine laboratory tests for hospitalized patients. Physicians-in-training will be cluster-randomized into two arms: (1) those who receive report cards (intervention group), (2) those who will not receive report cards (control group). We will study the use of routine laboratory tests over a pre-intervention period of 1 week and a post-randomization period of 1 week. We will study physician attitudes about the real-time feedback dashboard with qualitative assessments in focus groups after the completion of the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Any internal medicine physician-in-training scheduled to rotate through general medicine services at HUP during the study period will be included in the study.

Exclusion Criteria:

* Physicians-in-training pulled for weekend coverage or sick coverage will be excluded. Medical students will be excluded.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 154 (Actual)
Dates: Start 2015-12; Primary Completion 2016-06 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Routine laboratory tests/patient-day | 6 months
  the number of routine laboratory tests per patient-day ordered by the physicians-in-training

SECONDARY OUTCOMES:
Laboratory costs | 6 months
Routine imaging tests/patient-day | 6 months
Physicians' attitudes toward laboratory test use and receiving feedback | 6 months
  Focus groups

OTHER OUTCOMES:
Non-routine laboratory tests/patient-day | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Kira L Ryskina, MD, Principal Investigator — University of Pennsylvania

REFERENCES:
- [Background] Ryskina K, Jessica Dine C, Gitelman Y, Leri D, Patel M, Kurtzman G, Lin LY, Epstein AJ. Effect of Social Comparison Feedback on Laboratory Test Ordering for Hospitalized Patients: A Randomized Controlled Trial. J Gen Intern Med. 2018 Oct;33(10):1639-1645. doi: 10.1007/s11606-018-4482-y. Epub 2018 May 22. PMID 29790072
- [Result] Kurtzman G, Dine J, Epstein A, Gitelman Y, Leri D, Patel MS, Ryskina K. Internal Medicine Resident Engagement with a Laboratory Utilization Dashboard: Mixed Methods Study. J Hosp Med. 2017 Sep;12(9):743-746. doi: 10.12788/jhm.2811. PMID 28914280